CLINICAL TRIAL: NCT05499169
Title: Coach Pilot Study: Assessing Cognitive Function and Related Small Vessel Disease Markers After Intracerebral Hemorrhage; a Pilot Study
Brief Title: Coach Pilot Study: Assessing Cognitive Function and Related Small Vessel Disease Markers After Intracerebral Hemorrhage
Acronym: COACH
Status: Terminated | Type: Observational
Why Stopped: Did not meet recruitment target
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Marieke JH Wermer, MD, Professor, Leiden University Medical Center
Other Study IDs: P20.109
Record Dates: First submitted 2022-08-01; First posted 2022-08-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage; Hypertensive Hemorrhage, Intracranial; Cognitive Decline
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Hemorrhage; Intracranial Hemorrhage, Hypertensive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If participants give permission for Leiden University Medical Center (LUMC) Biobank sporadic cerebral amyloid angiopathy (sCAA) (part of the LUMC Biobank Neurological Diseases), an additional 50 ml blood will be drawn. These blood samples will be stored for future (yet unknown) biomarker analysis after approval of the participants. These blood samples will be handled confidentially and coded and will be stored in the LUMC Biobank sCAA Neurological Diseases. The regulations of the LUMC Biobank Neurological Diseases will be applicable to the LUMC Biobank sCAA under Neurological Diseases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 16 patients with CAA-related ICH: 16 patient above the age of 55 that fit the inclusion criteria. CAA-related ICH is defined as an ICH that meets the criteria for definite or probable CAA according to the Modified Boston Criteria.
- 16 patients with HA-related ICH: 16 patient above the age of 55 that fit the inclusion criteria. HA-related ICH is defined as ICH located in the basal ganglia, thalamus, or the deep white matter and the presence of hypertension defined as: on treatment for hypertension, or known with high blood pressure (two measurements systolic blood pressure (SBP) >140 or diastolic blood pressure (DBP) >90 mmHg) but not treated for hypertension.

SUMMARY:
The overall aim of this pilot study is to investigate the development of magnetic resonance imaging (MRI) and cerebrospinal fluid (CSF) markers after cerebral amyloid angiopathy (CAA)-related and hypertensive arteriopathy (HA)-related intracerebral hemorrhage (ICH) in relation to cognitive decline. The results from this pilot trial will be used to design a larger cohort study to investigate underlying mechanisms of cognitive decline after ICH. The study population consists of 32 patients; 16 patients with CAA-related ICH and 16 patients with HA-related ICH who are 55 years or older. Data will be collected at four measuring points: at baseline (during hospital admission for the ICH or at the outpatients clinic within one month of presentation with an acute ICH), after three months, after six months and after 12 months. Premorbid cognitive functioning will be assessed with the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) to select participants without pre-existing cognitive impairment.

DETAILED DESCRIPTION:
Dementia is a major contributor of dependence and disability in the ageing population and is mainly caused by neurodegenerative and cerebrovascular disease. Vascular cognitive impairment (VCI) occurs in at least 10% of patients who recover from an intracerebral hemorrhage (ICH) and has a major impact on post ICH recovery. In the acute phase of ICH, cognitive impairment may be caused directly by the hemorrhage damaging the brain parenchyma. In the chronic phase, however, further cognitive decline is also prevalent.

Cognitive decline after ICH might be caused by the underlying etiology of the ICH. The most frequent underlying small vessel diseases (SVD) that cause ICH are cerebral amyloid angiopathy (CAA) and hypertensive arteriopathy (HA). CAA and HA have their own radiological signatures of SVD markers which allow for in vivo tracking of disease progression using MRI. Although the initial clinical presentation these two types of SVD differs - CAA classically presents with a lobar ICH, whereas HA causes deep ICH - both groups of patients are at risk of developing dementia. However, it has recently been shown that patients with lobar ICH develop new onset dementia twice as often as patients with deep ICH. Whether underlying CAA pathology causes this increase, remains unclear. In addition, whether ICH accelerates the process of vascular damage and if cognitive decline can be predicted by certain disease markers is uncertain. Understanding the underlying mechanisms for cognitive decline after ICH helps to improve knowledge of prognosis and clinical management of patients who are recovering from ICH. The overall aim is to study cognitive decline in patients who recover from ICH and the relation with SVD markers. The results will be used to design a larger cohort study.

The study population are patients with ICH that have no family history of hereditary forms of ICH such as hereditary CAA (HCHWA-D) and no cognitive impairment before the ICH. Patients will be aged ≥ 55y, since the radiological Boston criteria for CAA-related ICH only include patients ≥ 55y. At baseline, the premorbid functional status will be assessed with the modified Rankin Scale (mRS) and Barthell index. A 3Tesla MRI will be performed to assess the most likely underlying cause of the ICH (patients with either CAA or HA-related ICH will be included). Stroke severity will be assessed with the National Institutes of Health Stroke Scale (NIHSS) and a neurologic exam will be performed. Participants will undergo an extensive interview on life-style, vascular risk factors and medication, and will undergo a blood withdrawal. Neuropsychological testing will be performed and questionnaires will be used for screening for depression, anxiety and psychopathology. In addition, participants will be asked to undergo a lumbar puncture to collect cerebrospinal fluid (CSF). After three months, neurological examination, and neuropsychological testing will be repeated. After six and 12 months, the neurological examination, the 3 Tesla MRI and neuropsychological testing will be repeated. Additionally, participants will be asked for a lumbar puncture at these two time points. The main parameters are cognitive decline (according to the neuropsychological assessment) at 12 months. Secondary outcomes are burden of SVD markers on MRI and CSF markers at baseline, at six months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55y
2. Ability and willingness to provide written informed consent.
3. Supratentorial ICH with CAA or HA as the most likely cause.

Exclusion Criteria:

1. Age < 55y
2. Unable to provide informed consent.
3. Pre-existing cognitive impairment assessed with the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE); scores between 53 - 63 reflect pre-existing cognitive impairment
4. Contra indications, such as: Contra-indications for 3T MRI. Examples of possible contra-indications are:

   * Claustrophobia
   * Pacemakers and defibrillators
   * Nerve stimulators
   * Intracranial clips
   * Intra-orbital or intraocular metallic fragments
   * Cochlear implants
   * Ferromagnetic implants
   * Hydrocephalus pump
   * Intra-uterine device
   * Permanent make-up
   * Tattoos above the shoulders
   * Reduced kidney function (estimated GFR < 30 ml/min/1,73m2; or nephrogenic systemic fibrosis / nephrogenic fibrosing nephropathy (NSF/NFD))
   * Known prior allergic reaction to gadolinium contrast or one of the constituents of its solution for administration

Contraindications for lumbar puncture:

* Intracranial tumor
* Compressio medullae
* Signs and symptoms of increased intracranial pressure
* Local infections of the skin
* A coagulopathy including use of anti-coagulant drugs (INR ≥ 1.8) or thrombocytopenia (<40)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patients with ICH that have no family history of hereditary forms of ICH such as hereditary CAA (HCHWA-D) and no cognitive impairment before the ICH. Patients will be aged ≥ 55y, since the radiological Boston criteria for CAA-related ICH only include patients ≥ 55y.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Cognitive decline (according to the neuropsychological assessment) | 12 months after ICH
  New onset cognitive impairment and dementia will be determined according to the Mini-Mental State Examination (MMSE) and compared between CAA-related and HA-related ICH.

SECONDARY OUTCOMES:
Burden of SVD markers on MRI markers at baseline, at six months and at 12 months | Baseline, at six months and at 12 months
  The presence and number of microbleeds (MBs), cortical superficial siderosis (cSS), white matter hyperintensities (WMH), chronic subarachnoid hemorrhage (cSAH), enlarged perivascular spaces (ePVS), microinfarcts, intragyral hemorrhages, cortical atrophy and other new and known small vessel biomarkers will be assessed on 3T and scored according to the STRIVE-criteria. These SVD markers will be added up to form a total MRI small vessel disease score. This total MRI small vessel disease score will be compared in patients at baseline, at six months and after twelve months.
Concentrations of p-tau181 in CSF at baseline, at six months and at 12 months | Baseline, at six months and at 12 months
  Concentrations of p-tau181 (in pg/ml) will be determined in the CSF of each patient at baseline, at six months and at 12 months. Changes in concentration will be calculated in each patient. Linear regression analysis will be used to examine associations of CSF markers primarily with the MMSE.
Concentrations of Aβ40 in CSF at baseline, at six months and at 12 months | At baseline, at six months and at 12 months
  Concentrations of Aβ40 (in pg/ml) will be determined in the CSF of each patient at baseline, at six months and at 12 months. Changes in concentration will be calculated in each patient. Linear regression analysis will be used to examine associations of CSF markers primarily with the MMSE.
Concentrations of Aβ42 in CSF at baseline, at six months and at 12 months | At baseline, at six months and at 12 months
  Concentrations of Aβ42 (in pg/ml) will be determined in the CSF of each patient at baseline, at six months and at 12 months. Changes in concentration will be calculated in each patient. Linear regression analysis will be used to examine associations of CSF markers primarily with the MMSE.
Concentrations of t-tau in CSF at baseline, at six months and at 12 months | At baseline, at six months and at 12 months
  Concentrations of t-tau will be determined in the CSF of each patient at baseline, at six months and at 12 months. Changes in concentration will be calculated in each patient. Linear regression analysis will be used to examine associations of CSF markers primarily with the MMSE.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis van Etten, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT05499169/Prot_000.pdf